CLINICAL TRIAL: NCT05614154
Title: Comparison of the Efficacy of Antiseptics With Povidone Iodine and Hypochlorous Acid Active Substance in Catheter Dressings in Preventing Central Catheter-Related Bloodstream Infection in Intensive Care Units
Brief Title: Comparison of the Efficacy of Antiseptics in Catheter Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vesile Eskici Ilgin, Vesile Eskici İlgin, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Vesile30
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: 3rd Level Intensive Care Unit
Keywords: central venous catheter; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Patients meeting the inclusion criteria Patients dressed with 1st group Povidone-iodine antiseptic (routinely applied antiseptic in the clinic)
Masking Description: Patients who met the criteria for participation in the study 2nd group patients dressed with antiseptic with hypochlorous active substance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone-iodine Group (Active Comparator): The care of patients with central venous catheters will be done with Povidone iodine as long as they stay in the intensive care unit
  Interventions: Other: hypochlorous active substance
- hypochlorous active substance (Experimental): The care of patients with central venous catheters will be done with antiseptic with hypochlorous active substance as long as they stay in the intensive care unit.
  Interventions: Other: hypochlorous active substance

INTERVENTIONS:
Other: hypochlorous active substance — Poviodin iyot

SUMMARY:
Intensive care units (ICUs) are care centers where many different technological tools and equipment are used to support the highest level of life functions for patients with severe physical condition. With the developing treatment and care methods, the use of more tools and equipment for invasive or non-invasive procedures has increased, however, complications related to the use of devices and the complications caused by them have also increased. Intensive care centers are centers where invasive procedures are frequently applied and instruments are used frequently, and central venous catheters (CVCs) are widely used, especially for patient-related reasons. CVCs have become one of the most important tools of intensive care units due to the different areas in which they are used and the benefits they provide.

DETAILED DESCRIPTION:
1.625 / 5.000 Çeviri sonuçları star_border A CVC is a cannula placed in a venous vein that goes directly to the heart. 4 CVCs are used for frequent blood sampling, continuous Total Parenteral Nutrition (TPN) administration, blood and blood product transfusions, hemodialysis, long-term fluid replacements, drug treatments in cases where vascular access cannot be used due to long-term and intensive treatments. It is used for a variety of purposes, such as the delivery of inotropes.

In addition to the benefits they provide, CVCs also have many negative side effects. The most common complications are infection, thrombosis and bleeding. central venous catheter-associated bloodstream infections (LVMI-CDE); It is seen as an important problem related to the use of central venous catheters in health services in ICUs.

The day the CVC is placed is recorded as day 1. Laboratory-confirmed BSI can be placed on the 3rd day of the catheter at the earliest, and the day after the catheter removal at the latest.9 The most important step in the management of LVMI-BSI is the prevention of infection. In order to prevent these unavoidable infections, precautions should be taken and antiseptic rules should be followed during the placement, use and maintenance of CVCs. Nurses are responsible for catheter care, monitoring and reporting in case of complications. Therefore, the specific care given by nurses has an effect on other catheter-related complications and increased infection. Catheter dressings can be considered as risk factors for bloodstream infection. For this reason, the antiseptics used during the dressing are also important.

Hypochlorous acid (HOCl), another antiseptic, is a highly effective product that is frequently used in dressings and wound care in recent years. Hypochlorous acid is also a physiological molecule synthesized by neutrophil cells during phagocytosis and plays an active role in the destruction of all microorganisms.

It has been shown in studies that HOCl inactivates various viruses, including coronaviruses, in less than 1 minute. 26 It has been stated that the use of HOCl in eyelid inflammation reduces the rate of bacteria on the skin surface. Twenty minutes after application of a saline hygiene solution containing HOCl at 100 ppm, more than 99% reduction in staphylococcal load was reported.27 In a clinical study of intraperitoneal wound care, in a randomized controlled study with forty-four patients aged 3-14 years, 20 patients were lavaged with 100 ml/kg isotonic into the peritoneal cavity and the wound was washed with 200 ml of isotonic, and 26 patients were poured 100 ml/kg into the peritoneal cavity. Lavage was done with HOCl and the wound was washed with 200 ml of HOCl. It was stated that no side effects were observed. HOCl is extremely ecological because its breakdown produces only brine and traces of chloride gas. It is economical as its source is only unsterilized tap water and salt.28 In a study examining the effect of stabilized hypochlorous acid solution (HOCl) on the killing rate, biofilm formation, antimicrobial activity in the biofilm on frequently isolated microorganisms and the migration rate of injured fibroblasts and keratinocytes, all microorganisms were killed within 0 minutes and the exact killing time was stated to be 12 seconds. The stabilized HOCl solution had dose-dependent positive effects on fibroblast and keratinocyte migration compared to povidone-iodine and medium alone. It was stated that it can be used as an ideal wound care agent.

In a study on diabetic foot wound, povidone iodine was compared with HOCl. The duration of antibiotic use decreased in cases where HOCl acid was used compared to povidone iodine. In the studies, in soft tissue and bone tissue; It has been shown to reduce inflammation and accelerate wound healing. Topically stabilized HOCl provides an optimal wound healing environment and when combined with silicone can be ideal for reducing scarring. Used as an antiseptic skin preparation, HOCl poses no concerns of ocular or ototoxicity. The fact that it is cheaper than other antiseptic solutions for dressings and is effective in many bacterial infections without damaging the tissue may cause more frequent use of hypochlorous acid. This study is extremely important in terms of providing evidence to the literature. Studies have shown that as a result of the correct nursing care and dressings made with the correct products, the rate of bloodstream infections, mortality and morbidity, as well as hospital costs due to the catheter, are greatly reduced. In this study, it was aimed to compare the effectiveness of antiseptics containing chlorhexidine, povidone iodine and hypochlorous acid active ingredient in catheter dressings in preventing central catheter-related bloodstream infection in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

1- 18 years or older 2- Opening the central venous catheter in the intensive care unit 3- Verbal consent from the relatives of the patients to participate in the study is accepted to participate in the study.

-

Exclusion Criteria:

1. Being under the age of 18
2. Exitus before the expected follow-up period of the patient
3. Being pregnant
4. Transferring from another unit or center to the Intensive Care Unit by CVC
5. Patients with a previous diagnosis of LVMI-CDE
6. Patients whose CVC was opened and CVC dressing was changed outside the control of the researcher -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
infection and viral signs tracking form | 4 times in 24 hours
  presence of infection in the central venous catheter site, if any, redness, temperature increase and presence of exudate around the catheter exit site, blood culture sampling date, body temperature/chills, number of blood cultures, microorganism name, vital signs (pulse, blood pressure, saturation, respiratory number) is included. Two blood cultures, peripheral and catheter, are taken as soon as the patient is placed in the catheter. In addition, if the patient has fever (> 38 °C), hypotension (systolic blood pressure < 90 mmHg) or oliguria (< 20 mL/hour) without any reason, and there is redness, swelling or purulent discharge around the catheter, the catheter blood culture is renewed.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile eskici İlgin, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No